CLINICAL TRIAL: NCT06673667
Title: A Phase 1, Randomized, Placebo-Controlled, First-in-Human, Single and Multiple Ascending Dose Study Designed to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Orally Administered KT-621 in Healthy Adult Participants
Brief Title: First-in-human Study of Orally Administered KT-621 in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kymera Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: KT621-HV-101
Record Dates: First submitted 2024-10-23; First posted 2024-11-05 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Healthy Participants Study
Keywords: Phase 1; STAT6; STAT6 degrader; targeted protein degrader

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The Sponsor is also masked to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- KT-621 (Active Comparator): Each participant receives either a single oral dose (SAD) or multiple oral doses (MAD) of KT-621.
  Interventions: Drug: KT-621
- Placebo (Placebo Comparator): Each participant receives either a single oral dose (SAD) or multiple oral doses (MAD) of matched placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KT-621 — Oral drug
  Arms: KT-621
Drug: Placebo — Oral drug
  Arms: Placebo

SUMMARY:
This is a first-in-human study to evaluate safety, pharmacokinetics, and pharmacodynamics of single and multiple dose levels of KT-621 in healthy male and female adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 19 to 55 years (inclusive) at the time of consent, with a weight of at least 50 kg if male or 40 kg if female, and a body mass index (BMI) between 18.0 and 30.0 kg/m² (inclusive) at Screening.
* Evidence of a personally signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study.
* Participants must be willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
* Male participants (and their partners of childbearing potential) and female participants must agree to the contraception requirements as specified in the clinical protocol.
* Female participants may not be pregnant, lactating, or breast-feeding or plan to become pregnant (including ova donation) within 30 days of last study drug administration.
* Female participants must have a negative result for pregnancy test at Screening and on admission to the CRU.

Exclusion Criteria:

* Participants who have a clinically relevant history of respiratory, gastrointestinal (GI), renal, hepatic, hematological, lymphatic, endocrinological, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, ophthalmological, or connective tissue diseases or disorders.
* Participants who have a clinically relevant surgical history (eg, surgery of the GI tract that could interfere with the PK of the trial medication) Note: prior appendectomy or cholecystectomy is not exclusionary.
* Participants with a history of alcohol or substance abuse within the previous 5 years.
* Participants who have any known factor, condition, or disease that might interfere with treatment compliance, study conduct or interpretation of the results such as drug or alcohol dependence or psychiatric disease.
* Participants who test positive for alcohol and drugs of abuse at Screening and on admission to the CRU.
* Participants who have acute GI symptoms at the time of Screening or admission to the CRU (eg, nausea, vomiting, diarrhea, heartburn).
* Participants whose results from clinical laboratory safety tests are outside the local reference range at Screening and on admission to the CRU.
* Participants who have previously received KT-621 in another cohort in this study.
* Participants who have been dosed with any investigational drug or device in a clinical study within 30 days or 5 half-lives (whichever is longer) of KT-621/placebo administration.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 118 (Actual)
Dates: Start 2024-10-22 (Actual); Primary Completion 2025-04-23 (Actual); Study Completion 2025-04-23 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | From enrollment through the safety follow-up visit on either Day 14 (SAD) or Day 38 (MAD)
Treatment-emergent potentially clinically-significant abnormalities in safety laboratory parameters: hematology | From enrollment through the safety follow-up visit on either Day 14 (SAD) or Day 38 (MAD)
  Hemoglobin, Hematocrit, Erythrocytes, Mean corpuscular volume, Platelets, Leukocytes, Eosinophils, Basophils Neutrophils Lymphocytes Monocytes
Treatment-emergent potentially clinically significant abnormalities in safety laboratory parameters: serum chemistry | From enrollment through the safety follow-up visit on either Day 14 (SAD) or Day 38 (MAD)
  Glucose, Blood urea nitrogen, Creatinine, Sodium, Potassium, Calcium, Chloride, Magnesium, Bicarbonate, Phosphate, Bilirubin, total and direct, Alkaline phosphatase, Aspartate transaminase (=SGOT), Alanine transaminase (=SGPT), Gamma glutamyl transferase, Total protein, Albumin, Creatine kinase, HbA1c, Lactate dehydrogenase (LDH)
Treatment-emergent potentially clinically significant abnormalities in safety laboratory parameters: coagulation | From enrollment through the safety follow-up visit on either Day 14 (SAD) or Day 38 (MAD)
  Activated partial thromboplastin time, Prothrombin time, International Normalized Ratio, Fibrinogen
Treatment-emergent potentially clinically significant abnormalities in electrocardiogram values: QTcF (milliseconds) | From enrollment through the safety follow-up visit on either Day 14 (SAD) or Day 38 (MAD)
Treatment-emergent potentially clinically significant abnormalities in vital signs: heart rate (beats per minute) | From enrollment through the safety follow-up visit on either Day 14 (SAD) or Day 38 (MAD)
Treatment-emergent potentially clinically significant abnormalities in vital signs: blood pressure (mmHg) | From enrollment through the safety follow-up visit on either Day 14 (SAD) or Day 38 (MAD)
Treatment-emergent potentially clinically significant abnormalities in vital signs: respiratory rate (breaths per minute) | From enrollment through the safety follow-up visit on either Day 14 (SAD) or Day 38 (MAD)
Treatment-emergent potentially clinically significant abnormalities in vital signs: temperature (degrees Celsius) | From enrollment through the safety follow-up visit on either Day 14 (SAD) or Day 38 (MAD)

SECONDARY OUTCOMES:
Maximum concentration (Cmax): observed maximum concentrations derived from plasma concentration data | Day 1 (SAD); Day 1, Day 7, and Day 14 (MAD)
Time to maximum concentration (Tmax): observed time to achieve maximum concentrations derived from plasma concentration data | Day 1 (SAD); Day 1, Day 7, and Day 14 (MAD)
Area under the curve (AUC0-last): Area under the plasma concentration-time curve calculated using non-compartmental analysis from time zero to the last observed timepoint | Day 1 (SAD); Day 1, Day 7, and Day 14 (MAD)
Area under the curve (AUC0-infinity): Area under the plasma concentration-time curve calculated using non-compartmental analysis from time zero to infinite time | Day 1 (SAD)
Area under the curve (AUC0-tau): Area under the plasma concentration-time curve calculated using non-compartmental analysis from time zero to end of the dosing interval | Day 1, Day 7, and Day 14 (MAD)
Terminal elimination half-life (t1/2): elimination half-life calculated using non-compartmental analysis | Day 1 (SAD) and Day 14 (MAD)
Fraction excreted: Fraction of drug excreted unchanged in urine | Day 14 (MAD)

OTHER OUTCOMES:
Change from baseline in STAT6 protein levels in whole blood and peripheral blood mononuclear cells (SAD) | Day 1
Change from baseline in STAT6 protein levels in whole blood, peripheral blood mononuclear cells, and skin (MAD) | Day 1 to Day 14

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Celerion, Phoenix, Arizona
  - Celerion, Lincoln, Nebraska

IPD SHARING:
Plan to Share IPD: No